CLINICAL TRIAL: NCT05958303
Title: Human Cerebral Blood Flow Regulation: Sex, Mechanism, and Stress Differences
Brief Title: HYPEROXIA Responses and ROS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2023-0850; 1R01HL150361-01 (NIH); EDUC/KINESIOLOGY (Other: UW Madison); Protocol Version 2/27/2024 (Other: UW Madison)
Record Dates: First submitted 2023-07-06; First posted 2023-07-24 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cerebrovascular Disorders
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antioxidant Cocktail (Experimental): The first dose will be 500 mg vitamin C, 200 IU vitamin E, and 300 mg of alpha lipoic acid 120 minutes before MRI. The second dose will be 500 mg vitamin C, 400 IU vitamin E, and 300 mg of alpha lipoic acid 60 minutes before MRI.
  Interventions: Dietary Supplement: Antioxidant Cocktail
- Placebo (Active Comparator): Placebo 120 minutes before MRI, followed by another dose of placebo 60 minutes before MRI.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Antioxidant Cocktail — Total dosing of 1000 mg vitamin C, 600 IU vitamin E, and 600 mg of alpha lipoic acid.
  Other Names: AOC
  Arms: Antioxidant Cocktail
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
30 participants (15 males and 15 females) who are ≥18 - ≤ 40 years old and considered healthy will be enrolled into this study to test the role of reactive oxygen species (ROS) in regulating cerebral blood flow (CBF). Participants can expect to be on study for 2 study visits over a 6 month period.

DETAILED DESCRIPTION:
Objective: The current objective is to determine whether biological sex influences CBF control in hyperoxia in healthy young adults without confounds of age or disease.

The investigators will address 3 specific questions:

1. Are cerebral vasoconstrictor responses to hyperoxia greater in men?
2. Do all brain regions respond equally, or are there regional differences-possibly varying by sex?
3. Do ROS regulate the decrease in CBF in a sex specific fashion?

This study will be conducted in compliance with federal investigational drug regulations (21 CFR 312) and Good Clinical Practice (GCP) guidelines, as well as state law and institutional policies.

Study Population: This study includes 30 total participants; (15 males and 15 females) who are ≥18 - ≤ 40 years old and considered healthy.

Approach: CBF testing will be performed in research-dedicated MRI systems on UW campus. Participants will experience normoxia followed by hyperoxia conditions during each of the 2 study visits. Study design focuses on the use of an acute oral antioxidant cocktail (AOC) to test ROS signaling as a potential mechanism explaining sex differences in CBF control. To do this, 2 MRI visits in a double-blind placebo-controlled design will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age between ≥18 - ≤40 years

Exclusion Criteria:

* Hypertensive

  * >125 mmHg systolic blood pressure; or
  * >80 mmHg diastolic blood pressure
* BMI ≥25 kg/m2
* Fasting blood glucose ≥100 mg/dl
* LDL cholesterol ≥130 mg/dl
* Triglycerides ≥150 mg/dl
* Current diagnosis or history of:

  * peripheral vascular disease
  * hepatic disease
  * renal disease
  * lung disease
  * gastrointestinal disorders/bleeding
  * hematologic disease
  * stroke
  * myocardial infarction
  * coronary heart disease
  * congestive heart failure
  * heart surgery
  * prediabetes
  * diabetes mellitus (type 1, type 2, MODY, or others)
  * sleep apnea
  * hypertension
  * some autoimmune diseases, such as inflammatory bowel disease or systemic lupus erythematosus (exclusion at discretion of reviewing MD)
* Current smoking, defined as the use of tobacco or nicotine products >5 times in the past 30 days.
* Cardiovascular medication use
* NSAID sensitivity
* Any contraindications of having an MRI

  o (e.g. the requirement of anxiolytics in order to complete an MRI scan)
* Irregular menstrual cycle (females only)
* Medical conditions that can affect the menstrual cycle, such as hyperprolactinemia, prolactinoma, hypercortisolemia, and congenital adrenal hyperplasia (females only)
* Pregnancy, breast feeding, or plans to conceive within the next 3 months (females only)
* Polycystic ovary syndrome (females only)
* Hirsutism defined as unwanted and/or excessive hair growth on the face, chest, or back (females only)
* Levonorgestrel intrauterine device (IUD) (females only)
* Hormonal birth control will not be allowed in women, in order to control for high variability between type, dose, and route of therapy. However, in discussion with Dr. Davis (Co-I) and Dr. Laura Cooney M.D., physician experts in medical and reproductive endocrinology and infertility, there are two broad exceptions to this birth control criteria:

  1. Copper intrauterine devices (IUDs) will be allowed as they do not change systemic sex hormone levels).
  2. Women currently taking hormonal birth control (i.e. contraceptive pills, patch, ring) for contraception only (not for a medical condition such as those listed in exclusion criteria above) may consider temporarily stopping to become eligible for enrollment. Hormonal birth control must be stopped at least one month prior to Study Visit 1 to provide time for menstruation to resume. Then stoppage continues through the last planned study visit. Screening information will be reviewed by endocrinology physicians to determine eligibility and timing on this issue (details below).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Cerebral Blood Flow: Normoxia | up to 6 months
  Participants will be randomized to AOC or placebo. Normoxia measures will be collected under each condition in the MRI over 2 study visits.
Cerebral Blood Flow: Hyperoxia | up to 6 months
  Participants will be randomized to AOC or placebo. Hyperoxia measures will be collected under each condition in the MRI over 2 study visits.

CONTACTS AND LOCATIONS:
Overall Officials: William G Schrage, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No